CLINICAL TRIAL: NCT02832388
Title: Primary Aldosteronism: a Study of Diagnostic Approach and Treatment Outcome in Western Norway
Brief Title: Primary Aldosteronism in Western Norway
Status: Recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Oslo University Hospital (Other); Helse Stavanger HF (Other Government); Helse Fonna (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/742
Record Dates: First submitted 2016-01-25; First posted 2016-07-14 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hyperaldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples are collected from each study participants for routine biochemistry and for biopanning. Additional saliva and hair samples may be sampled.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Primary aldosteronism patients for cardiac MRI: A subgroup of primary aldosteronism (PA) patients perform a cardiac MRI, including stress-testing with adenosine, and are compared to a sex- and age-matched group of healthy controls who perform the same MRI procedure
- Healthy controls: Healthy controls that are age-and sex-matched to the subgroup of PA patients performing cardiac MRI, perform MRI including adenosine as stress-test.
- Primary aldosteronism patients diagnosed from 2013 onwards: All PA patients diagnosed or subtyped at Haukeland University from 2013 onwards are asked for inclusion in the main observational PA-study.
  From 2025 onwards, PA patients diagnosed or subtyped at Oslo University hospital will also be included.

SUMMARY:
In this study the investigators aim to identify and include consecutively patients with primary aldosteronism (PA) diagnosed in the Western and Mid-parts of Norway, to describe the characteristics of these patients, to explore the cardiac effects of PA before and after specific treatment, and to identify long-term outcomes after treatment. One subgroup of the PA patients perform echocardiography to assess left ventricular systolic myocardial function before and after treatment. One subgroup of PA patients perform cardiac MRI to assess myocardial mass, myocardial fibrosis and myocardial function in rest and during stress, before and after treatment. For the cardiac MRI substudy, the PA patients are compared with a group of healthy controls, also included in the study.

From 2022 onwards, PA patients diagnosed or subtyped with adrenal vein sampling at Oslo University Hospital will additionally be included in the study, thereby providing a national registration of PA patients.

DETAILED DESCRIPTION:
From June 2013, all newly diagnosed patients with primary aldosteronism (PA) either diagnosed at Haukeland University Hospital (HUS) or admitted to HUS for subtype testing with adrenal vein sampling, have been asked for inclusion in the study. All included patients have a base-line study visit where clinical information is registered, and baseline blood and urine samples are collected. Echocardiography will be performed in a subgroup of patients before and 1 year after start of specific PA treatment. After start of definite medical or surgical treatment the patients are followed up with regularly new study visits. From 2025 onwards, PA patients diagnosed or subtyped with adrenal vein sampling at Oslo University Hospital will additionally be included in the study, thereby providing a national registration of PA patients.

A subgroup of the included PA study patients also perform a Cardiac MRI. Cine-MRI, velocity-encoded MRI, MRI images during continuous adenosine infusion and MRI images after gadolinium contrast injection are performed, and compared to a group of age- and sex-matched healthy controls.

From 2025 onwards, PA patients either diagnosed or performing subtyping with adrenal vein sampling at Oslo University Hospital will likewise be asked for study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis or strong suspicion of primary aldosteronism
* Age 18-85

Exclusion Criteria:

* Active cancer disease at time of inclusion

Exclusion criteria for subgroup of primary aldosteronism-patients and healthy controls who perform cardiac MRI:

* Asthma/chronic obstructive pulmonary disease ,
* Use of dipyridamole
* Claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with primary aldosteronism diagnosed or subtyped at Haukeland University hospital from 2013 onwards. From Autumn 2020 onwards, patients diagnosed or subtyped at Oslo University Hospital are additionally included.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Long-term clinical outcome after surgical and medical treatment of PA | 5 years
  Systolic and diastolic blood pressure (mm Hg) will be measured after specific PA treatment for estimation of clinical blood pressure outcome. In adrenalectomized patients clinical outcome will be determined following the international standardized Primary Aldosteronism Surgery Outcome (= PASO) criteria.
Long-term biochemical outcome after surgical treatment of PA | 5 years
  Biochemical outcome after unilateral adrenalectomy will be determined by measurement of aldosterone (pmol/L), direct renin-concentration (mIE/L) for estimation of aldosterone/renin-ratio and potassium (mmol/L) in blood, following the international standardized PASO (primary aldosteronism surgery outcome) criteria.

SECONDARY OUTCOMES:
Echocardiographic assessment of left ventricular mass in PA patients before and after treatment | 3 years
  Echocardiography is applied to assess the rate of increased left ventricular mass (g/m2.7 )before and after specific PA treatment. Data will be compared with a control group of patients with primary hypertension (HT), participating in the FAT-associated CardiOvasculaR dysfunction (FATCOR) study, which is a study cohort established at the European Society of Hypertension Excellence Centre in Bergen.
Echocardiographic assessment of left ventricular systolic function measured as global longitudinal strain in PA patients before and after treatment | 3 years
  Echocardiography is applied to assess the rate of reduced left ventricular systolic myocardial function assessed as global longitudinal strain, before and after specific PA treatment. Data will be compared with a control group of primary hypertension participating in the FAT-associated CardiOvasculaR dysfunction (FATCOR) study, which is a study cohort established at the European Society of Hypertension Excellence Centre in Bergen.
Echocardiographic assessment of left ventricular systolic function measured as midwall shortening in PA patients before and after treatment | 3 years
  Echocardiography is applied to assess the rate of reduced left ventricular systolic myocardial function before and after specific PA treatment, measured as midwall shortening (%). Data will be compared with a control group of primary hypertension participating in the FAT-associated CardiOvasculaR dysfunction (FATCOR) study, which is a study cohort established at the European Society of Hypertension Excellence Centre in Bergen.
Incidence of reduced quality of life in PA patients before and after treatment, assessed by Short Form Health Surveys (SF-36/RAND-36) | 5 years
  Quality of life is measured in PA patients before, 1 year and 5 years after specific PA treatment, measured by the approved quality of life Short Form Health Surveys SF-36 and RAND-36, to detect the incidence of reduced quality of life compared with results from the healthy population. SF-36 was used in the period 2013-2016, and has from 2016 onwards been replaced by RAND-36.
Cardiac MRI assessment of left ventricular mass in PA patients before and after treatment | 3 years
  Cardiac MRI is performed to assess change of left ventricular mass after specific PA treatment
Cardiac MRI assessment of myocardial fibrosis in PA patients compared with healthy controls | 3 years
  Cardiac MRI with T1 mapping is performed to assess the presence of cardiac fibrosis in PA patients before and after specific PA treatment, compared with a control group of healthy controls
Cardiac MRI assessment of left coronary flow reserve | 3 years
  Stress testing during cardiac MRI is performed in PA patients and a control group of healthy controls to assess the rate of reduced coronary flow reserve in PA patients before and after specific PA treatment, compared with a control group of healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne A Grytaas, MD PhD, Principal Investigator — Haukeland University Hospital; Anders P Jørgensen, MD PhD, Study Director — Oslo University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Oslo University Hospital, Oslo

IPD SHARING:
Plan to Share IPD: No